CLINICAL TRIAL: NCT03179241
Title: SDR-Auswertung, Unterteil Kognition, Bildgebung, Lebensqualität
Brief Title: Outcome After Selective Dorsal Rhizothomy Concerning Life Quality, Cerebral Imaging and Cognition
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Anne van Riesen, MD, Charite University, Berlin, Germany
Other Study IDs: SDR-KoBL
Record Dates: First submitted 2017-06-05; First posted 2017-06-07 (Actual); Last update posted 2018-07-19 (Actual); Status verified 2018-07

CONDITIONS: Cerebral Palsy, Spastic
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Selektive dorsal rhizotomy (SDR) has been used as treatment option in children suffering from cerebral palsy (CP) for several decades and multiple studies demonstrated its benefits. Nevertheless, there are still no proven strategies for patient selection, optimal point of time for the operation or pre- and postoperative therapies. The evaluation of the impact of selective motor control, cognition and cerebral imaging findings on the motor outcome and life quality in children with CP who underwent SDR at the Charité University clinics will clarify these critical points in daily care for patients with CP.

DETAILED DESCRIPTION:
SDR at the Charité University clinics. Two study visits before surgery and during the follow-up 3 months, 6 months, 12 months, 24 months and 5 years post-operatively.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of cerebral palsy
* able to perform most tasks according to study protocols
* parents and physician decided to perform SDR

Exclusion Criteria:

* not able to perform any tasks according to study protocols
* no candidate for SDR

Ages: 2 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All patients treated with SDR at the Charité University clinics and who are able to perform tasks according to study protocols are eligible to enroll.
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2017-10-14 (Actual); Primary Completion 2021-10-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
Motor function measured by GMFCS | 5 years
  Ability of a child to perform specified motor tasks, measured by GMFCS and GMFM-88
Motor function measured by GMFM-88 | 5 years
  Ability of a child to perform specified motor tasks, measured by GMFCS and GMFM-88

SECONDARY OUTCOMES:
Quality of life measured by "Disabkids"-Questionaire (German version) | 5 years
  Measured by "Disabkids"-Questionaire (German version) and "kid screen"
Quality of life measured by questionaire "kid screen" | 5 years
  Measured by "kid screen"
Selective motor control | 5 years
  Measured by SCALE (Fowler et al., 2009)
Spasticity by modified Ashworth scale | 5 years
  Measured by modified Ashworth scale and Tardieu scale
Spasticity by modified Tardieu scale | 5 years
  Measured by modified Ashworth scale and Tardieu scale
Contractures by range of motion (ROM) | 5 years
  Measured by range of motion (ROM)

CONTACTS AND LOCATIONS:
Overall Officials: Anne K van Riesen, M.D., Principal Investigator — social pediatric center, departement of neuropediatrics
Locations (1):
- Charité University clinics, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No